CLINICAL TRIAL: NCT05745714
Title: International Proof of Concept Therapeutic Stratification Trial of Molecular Anomalies in Relapsed or Refractory HEMatological Malignancies in Children, Subprotocol C Ruxolitinib + Venetoclax + Dexamethasone + Cyclophosphamide and Cytarabine in Pediatric Patients With Relapsed or Refractory Hematological Malignancies
Brief Title: HEM-iSMART-C: Ruxolitinib + Venetoclax + Dexamethasone + Cyclophosphamide and Cytarabine in Pediatric Patients With Relapsed or Refractory Hematological Malignancies
Acronym: HEM-iSMART C
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Princess Maxima Center for Pediatric Oncology (Other)
Collaborators: Innovative Therapies For Children with Cancer Consortium (Other); IBFM (Industry); Fight Kids Cancer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-501867-42-00
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Acute Lymphoblastic Leukemia, in Relapse; Lymphoblastic Lymphoma (Precursor B-Lymphoblastic Lymphoma/Leukaemia) Recurrent; Lymphoblastic Lymphoma (Precursor T-Lymphoblastic Lymphoma/Leukaemia) Recurrent; Lymphoblastic Lymphoma (Precursor B-Lymphoblastic Lymphoma/Leukaemia) Refractory; Lymphoblastic Lymphoma (Precursor T-Lymphoblastic Lymphoma/Leukaemia) Refractory
Keywords: acute lymphoblastic leukemia; Lymphoblastic lymphoma; Biomarker driven clinical trial; Ruxolitinib; Venetoclax; Chemotherapy; Relapse; Children; Adolescents; Young adults
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Recurrence; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — ruxolitinib; venetoclax; Dexamethasone; Cyclophosphamide; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib + venetoclax + dexamethasone + cyclophosphamide + cytarabine (Experimental): Each cycle has 28 days
  Cycle 1: All patients will receive 14 days of of ruxolitinib (days 1-14), 28 days of venetoclax (days 1-28), one block of five days of dexamethasone (days 1-5), one dose of cyclophosphamide (day 3) and two blocks of four consecutive days of cytarabine (days 5 to 8 and days 12 to 15). A 1-day venetoclax ramp-up is proposed in this study.
  Cycle 2 and subsequent cycles:
  All patients will receive 14 days of of ruxolitinib (days 1-14), 28 days of venetoclax (days 1-28), one block of five days of dexamethasone (days 1-5), one dose of cyclophosphamide (day 1) and two blocks of four consecutive days of cytarabine (days 3 to 6 and days 10 to 13).
  Patients in dose level -1, will receive a lower dose of venetoclax compared to dose level 1.
  Patients in dose level 2, will receive a higher dose of venetoclax compared to dose level 1.
  All patients receive age adapted intrathecal chemotherapy.
  Interventions: Drug: Ruxolitinib; Drug: Venetoclax; Drug: Dexamethasone; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: intrathecal chemotherapy

INTERVENTIONS:
Drug: Ruxolitinib — oral
Drug: Venetoclax — oral
Drug: Dexamethasone — oral/intravenous
Drug: Cyclophosphamide — intravenous
Drug: Cytarabine — intravenous
Drug: intrathecal chemotherapy — IT: Methotrexate +/- prednisone/hydrocortisone/cytarabine according to the degree of central nervous involvement

SUMMARY:
HEM-iSMART is a master protocol which investigates multiple investigational medicinal products in children, adolescents and young adults (AYA) with relapsed/refractory (R/R) ALL and LBL. Sub-protocol C is a phase I/II trial evaluating the safety and efficacy of ruxolitinib and venetoclax in combination with dexamethasone, cyclophosphamide and cytarabine in children and AYA with R/R ped ALL/LBL whose tumor present with alterations in the IL7R/JAK-STAT pathway.

DETAILED DESCRIPTION:
HEM-iSMART is a master protocol with sub-protocols. The overarching objective is that introducing targeted therapy using a biomarker driven approach for treatment stratification may improve the outcome of children with R/R acute lymphoblastic leukemia (ALL) and lymphoblastic lymphoma (LBL) It is characterized by a shared framework that allows for the investigation of multiple IMPs and generate pivotal safety and efficacy evidence within the sub-protocols to establish and define the benefits and risks of new treatments for children with R/R leukemia.

Sub-Protocol C within HEM-iSMART, is a phase I/II, multicenter, international, open-label clinical trial designed to evaluate the safety, tolerability, pharmacokinetics (PK) and efficacy of ruxolitinib with venetoclax in combination with dexamethasone, cyclophosphamide and cytarabine in children, adolescents and young with R/R ALL and LBL. Patients with alterations in the IL-7R and/or JAK-STAT signaling pathways will be eligible for sub-protocol C.

ELIGIBILITY:
Inclusion Criteria:

1. Children between 1 year (≥ 12 months) and 18 years of age at the time of first diagnosis and less than 21 years at the time of inclusion
2. Performance status: Karnofsky performance status (for patients >12 years of age) or Lansky Play score (for patients ≤12 years of age) ≥ 50% (Appendix I).
3. Written informed consent from parents/legal representative, patient, and age-appropriate assent before any study specific screening procedures are conducted, according to local, regional or national guidelines.
4. Patients must have had advanced molecular profiling and flow-cytometric analysis of their recurrent or refractory disease at a time-point before the first inclusion into this trial (see section 9.1 for detailed description of the molecular diagnostics required). Drug response profiling and methylation is highly recommended but not mandatory. Patients with molecular profiling at first diagnosis lacking molecular diagnostics at relapse or refractory disease may be allowed to be included after discussion with the sponsor.
5. Patients whose tumor presents alterations in the IL-7R and/or JAK-STAT signaling pathways including but not limited to the following are eligible: CRLF2: Rearrangements and mutations leading to CRLF2 overexpression (P2RY8-CRLF2, IGH-CRLF2, and CRLF2 F232C), CRFL2 overexpression; EPOR: Truncating rearrangements or mutations in exon 8, EPOR fusions; JAK1/2/3: Recurrent or novel missense and in-frame indel mutations in or flanking the pseudokinase and kinase domains, JAK fusion; IL7R: Recurrent or novel missense or in-frame indel mutations in the transmembrane domain; SH2B3: Copy number deletions, or mutations that result in frameshifts or premature termination; JAK2: In frame fusions retaining the tyrosine kinase domain; USP9X truncating mutation or USP9X-DDX3X fusion; STAT5B and DNM2 mutations; PTPN2 deletion described as involved in IL7R/JAK/STAT pathway activation; IL7R mutations
6. Adequate organ function:

   * RENAL AND HEPATIC FUNCTION (Assessed within 48 hours prior to C1D1) :

     * Serum creatinine ≤ 1.5 x upper limit of normal (ULN) for age or calculated creatinine clearance as per the Schwartz formula or radioisotope glomerular filtration rate ≥ 60 mL/min/1.73 m2.
     * Direct bilirubin ≤ 2 x ULN (≤ 3.0 × ULN for patients with Gilbert's syndrome).
     * Alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) ≤ 5 x ULN; aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase/SGOT ≤ 5 x ULN. Note: Patients with hepatic disfunction related to the underling disease can be eligible even if they do not fulfill the aforementioned values for hepatic transaminases. In these cases, patients need to be discussed with the sponsor to confirm the eligibility.
   * CARDIAC FUNCTION:

     * Shortening fraction (SF) >29% (>35% for children < 3 years) and/or left ventricular ejection fraction (LVEF) ≥50% at baseline, as determined by echocardiography or MUGA.
     * Absence of QTcF prolongation (QTc prolongation is defined as >450 msec on baseline ECG, using the Friedericia correction), or other clinically significant ventricular or atrial arrhythmia.

   Exclusion Criteria:
7. Pregnancy or positive pregnancy test (urine or serum) in females of childbearing potential. Pregnancy test must be performed within 7 days prior to C1D1.
8. Sexually active participants not willing to use highly effective contraceptive method (pearl index <1) as defined in CTFG HMA 2020 (Appendix II) during trial participation and until 6 months after end of antileukemic therapy.
9. Breast feeding.
10. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter drug absorption of oral drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, or malabsorption syndrome) in case of oral IMPs.
11. Patients whose tumor present known mutationts confering resistance to JAK inhibitors: JAK1 Phe958 and Pro960 mutations and JAK2 Y931C mutations.
12. Patients whose tumor present known mutationts confering resistance to venetoclax (e.g. BCL2 mutations of venetoclax binding-site (Gly101Val mutation, Phe104Leu/Cys mutations).
13. Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to the study drugs, or drugs chemically related to study treatment or excipients that contraindicate their participation, including conventional chemotherapeutics (i.e. cytarabine and cyclophosphamide when applicable, intrathecal agents) and corticoids.
14. Known active viral hepatitis or known human immunodeficiency virus (HIV) infection or any other uncontrolled infection.
15. Severe concomitant disease that does not allow treatment according to the protocol at the investigator's discretion.
16. Subjects unwilling or unable to comply with the study procedures.
17. Previous treatment with ruxolitinib and venetoclax in combination (Patients who have previously received any of these two drugs separately can be eligible for this sub-protocol).
18. Current use of a prohibited medication or herbal preparation or requires any of these medications during the study. See Section 7, Appendix III and IV for details. In general, CYP3A4 inhibitors/Pgp inhibitors, moderate or strong inducers of CYP3A4 or drugs inducing QTc changes (prolongation of the QT interval or inducing Torsade de Points) are not permitted. Among others and not exclusively that relates to antiviral, antifungal, antibiotic, antimalarial, antipsychotic and antidepressive drugs.
19. Patients who have consumed grapefruit, grapefruit products, Seville oranges (Including marmalade containing Seville oranges) or starfruit within 72 hours prior to the first dose of study drug.
20. Unresolved toxicity greater than NCI CTCAE v 5.0 ≥ grade 2 from previous anti-cancer therapy, including major surgery, except those that in the opinion of the investigator are not clinically relevant given the known safety/toxicity profile of the study treatment (e.g., alopecia and/or peripheral neuropathy related to platinum or vinca alkaloid based chemotherapy) (Common Terminology Criteria for Adverse Events (CTCAE) (cancer.gov).
21. Active acute graft versus host disease (GvHD) of any grade or chronic GvHD of grade 2 or higher. Patients receiving any agent to treat or prevent GvHD post bone marrow transplant are not eligible for this trial.
22. Received immunosuppression post allogenic HSCT within one moth of study entry.
23. History of bone disorders such as osteogenesis imperfecta, rickets, renal osteodystrophy, osteomyelitis, osteopenia, fibrous dysplasia, osteomalacia etc. prior to the underlying diagnosis.
24. History of progressive multifocal leuko-encephalopathy (PML).
25. History of endocrine or kidney related growth retardation prior to the underlying diagnosis.
26. Evidence of clinically active tuberculosis (clinical diagnosis per local practice).
27. Wash-out periods of prior medication:

    1. CHEMOTHERAPY: At least 7 days must have elapsed since the completion of cytotoxic therapy, with the exception of hydroxyurea, 6-mercaptopurine, oral methotrexate and steroids which are permitted up until 48 hours prior to initiating protocol therapy. Patients may have received intrathecal therapy (IT) at any time prior to study entry.
    2. RADIOTHERAPY: Radiotherapy (non-palliative) within 21 days prior to the first dose of drug. Palliative radiation in past 21 days is allowed.
    3. HEMATOPOIETIC STEM CELL TRANSPLANTATION (HSCT):

       * Autologous HSCT within 2 months prior to the first study drug dose.
       * Allogeneic HSCT within 3 months prior to the first study drug dose.
    4. IMMUNOTHERAPY: At least 42 days must have elapsed after the completion of any type of immunotherapy other than monoclonal antibodies (e.g. CAR-T therapy)
    5. MONOCLONAL ANTIBODIES AND INVESTIGATIONAL DRUGS: At least 21 days or 5 times the half-life (whichever is shorter) from prior treatment with monoclonal antibodies or any investigational drug under investigation must have elapsed before the first study drug.
    6. SURGERY: Major surgery within 21 days of the first dose. Gastrostomy, ventriculo-peritoneal shunt, endoscopic ventriculostomy, tumor biopsy and insertion of central venous access devices are not considered major surgery.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2032-02-01 (Estimated); Study Completion 2032-02-02 (Estimated)

PRIMARY OUTCOMES:
Phase I: Maximum tolerated dose (MTD) / Recommended phase 2 dose (RP2D) | 3 years
  Defined as the highest dose level tested at which 0/6 or 1/6 patients experiences dose limiting toxicities (DLT) during course 1 with at least 2 patients experiencing DLT at the next higher dose
Phase II: Best Overall Response Rate (ORR) | 6 years
  For patients with leukemia: CR and MRD response after 1 cycle of treatment. This includes determination of CR, CRp, CRi and minimal residual disease (MRD) negativity rate in patients suffering from overt morphological relapse of T-ALL at time of enrolment (morphological disease (M2/M3)), and the MRD negativity rate in those that entered with high-MRD levels but in morphological CR. These results will together be presented as a composite endpoint Overall Response rate (ORR). MRD negativity will be defined as ≤1x10-4 as generated by multi-parameter flow cytometry.
  For patients with lymphoma: Response in LBL patients is defined as CR, PR, minor response (MR) as defined in International pediatric NHL response criteria. In case of bone-marrow involvement MRD will be taken into account.
  For patients with lymphoma: Response in LBL patients is defined as CR, PR, minor response (MR) as defined in International pediatric NHL response criteria.

SECONDARY OUTCOMES:
Overall survival (OS) | 7 years
  Defined as time from C1D1 until death of any cause.
Event-free survival (EFS) | 7 years
  Defined as time from C1D1 to the first event (subsequent relapse after CR (including molecular reappearance), death of any cause, failure to achieve remission (CR, CRp or CRi), or secondary malignancy).
Cumulative incidence of relapse (CIR) | 7 years
  Estimate of the risk, that a patient will develop a relapse over a specified period of time.
Number of patients proceeding to hematopoietic stem cell transplantation (HSCT) after the experimental therapy | 7 years
  The rate of those proceeding to subsequent allogenic HSCT
Cumulative overall response rate (ORR) | 7 years
  Defined as the CR, CRp, CRi and MRD negativity rates after more than 1 cycle of treatment.
Rate of dose limiting toxicities (DLTs) | 7 years
  Number of participants with dose limiting toxicities (DLTs).
Peak plasma concentration (Cmax) | 6 years
  Estimation of ruxolitinib Cmax.
Peak plasma concentration (Cmax) | 6 years
  Estimation of venetoclax Cmax.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Zwaan, Prof. Dr., Study Chair — Princess Máxima Center; Paco Bautista, MD PhD, Principal Investigator — Princess Máxima Center
Locations (33):
- St. Anna Kinderspital, Vienna, Austria
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Rigshospitalet Copenhagen, Copenhagen, Denmark
- Helsinki University Hospital, New Children's Hospital, Helsinki, Finland
- France (6):
  - Hôpital des Enfants GH Pellegrin - CHU de Bordeaux, Bordeaux
  - CHRU Lille - Hôpital Jeanne de Flandre, Lille
  - Centre Léon Bérard, Lyon
  - Hopital La Timone - Enfants, Marseille
  - CHU Nantes Hôpital Mère-Enfant, Nantes
  - Hôpital Robert Debré, Paris
- Germany (5):
  - Universitätsklinikum Augsburg, Augsburg
  - Charité Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Münster, Münster
- Our Lady's Hospital for Sick Children, Dublin, Ireland
- Israel (2):
  - Schneider's Children's Medical Center, Petah Tikva
  - Sheba Medical Center Hospital, Ramat Gan
- Italy (5):
  - IRCCS Istituto Giannina Gaslini, Genova
  - Fondazione MBBM c/o Centro ML Verga, Monza
  - Padova Azienda Ospedaliera, Padua
  - Ospedale Pediatrico Bambino Gesù, IRCCS, Roma
  - Ospedale Infantile Regina Margherita, Turin
- Princess Máxima Center for Pediatric Oncology, Utrecht, Utrecht, Netherlands
- Oslo University Hospital, Oslo, Norway
- Spain (3):
  - Hospital Sant Joan de Déu de Barcelona, Barcelona
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - La Fe, Valencia
- Karolinska university hospital, Stockholm, Sweden
- United Kingdom (4):
  - Bristol Royal Hospital for Children, Bristol
  - Great Ormond Street Hospital for Children NHS Trust, London
  - Great North Children's Hospital, Newcastle
  - Royal Marsden NHS Trust, Sutton

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data will be used to generate a publication.
Supporting Information: CSR
Time Frame: SRs will also be provided at the end of specific sub-protocols or specific phases of a sub-protocol, and when needed for regulatory purposes.
  Examples for generating 'primary CSRs' may include:
  * After Last Patient Last Visit (LPLV) in a study having ORR as endpoint.
  * After the RP2D is determined in a Phase I part of a given sub-protocol.
  * After the follow-up of a specific sub-protocol is completed.
Access Criteria: A summary of the study results will be made public via clinicaltrials.gov as well as to Ethical committees/ Health Authorities and all participating patients by providing them through their treating physicians a patient letter with a summary of the results.